CLINICAL TRIAL: NCT01068015
Title: A COMMUNITY-BASED, RANDOMIZED CONTROLLED TRIAL TO EVALUATE THE EFFICACY OF COMPREHENSIVE HIV/STIs INTERVENTION AMONG MEN WHO HAVE SEX WITH MEN IN 8 CITIES IN CHINA
Brief Title: (Men Who Have Sex With Men) MSM Community Intervention Trial
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Center for AIDS/STD Control and Prevention, China CDC (Other Government)
Collaborators: Yunnan Center for Disease Control and Prevention (Other); Xinjiang Center for Disease Control and Prevention (Other); Sichuan Center for Disease Control and Prevention (Other Government); Guangxi Center for Disease Control and Prevention (Other Government); Guizhou Center for Disease Control and Prevention (Other); Shanghai Center for Disease Control and Prevention (Other); Beijing Center for Disease Control and Prevention (Other Government); Chongqing Center for Disease Control and Prevention (Other)
Responsible Party: Professor Zunyou Wu, National Center for AIDS/STD Control and Prevention, China CDC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Intervention20100105
Record Dates: First submitted 2010-02-11; First posted 2010-02-12 (Estimated); Last update posted 2010-04-08 (Estimated); Status verified 2010-04

CONDITIONS: HIV; Syphilis; Herpesvirus 2, Human
Keywords: MSM; Intervention; Popular Opinion Leader; Male Circumcision; HIV; Syphilis; HSV-2
MeSH Terms: conditions — Syphilis | interventions — Circumcision, Male

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): This arm receives free circumcision service, POL intervention, intensive HIV counseling and intensive condom promotion.
  Interventions: Other: behavior intervention and male circumcision
- usual (No Intervention): This arm receives no extra HIV prevention services.
  Interventions: Other: behavior intervention and male circumcision

INTERVENTIONS:
Other: behavior intervention and male circumcision — MSM in intervention arm can receive circumcision service for free, POL intervention, intensive HIV counseling and intensive condom promotion.

SUMMARY:
The purpose of this study is to evaluate the effectiveness of the community based comprehensive HIV/STIs intervention among MSMs in China.

DETAILED DESCRIPTION:
National sentinel surveillance data show that HIV infections are increasing fast among men who have sex with men(MSM) in China. In some cities HIV prevalence among MSM is higher than 10%.It is urgent for China to explore innovative intervention to reduce HIV/AIDS transmission among this population.

The purposes of this study are:

1. To evaluate the effectiveness of comprehensive interventions to decrease the HIV/STIs incidence among MSM population in China. The comprehensive intervention components include male circumcision, POL intervention, HIV testing and counseling and condom promotion.
2. To determine the acceptability of male circumcision among MSM population in China.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or above
* Male have oral sex or anal sex within 6 months with a man
* Accept questionnaire survey and blood test
* Can participate in three surveys in one year
* HIV Negative
* No mental disease and can understand informed consent

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3214 (Actual)
Dates: Start 2009-06; Primary Completion 2010-11 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
HIV incidence | March 1,2010 to Dec,31,2010

SECONDARY OUTCOMES:
Syphilis, HSV-2 incidence | 1,Mar.,2009 to 31,Dec,2010
Frequency of condom uses, number of sexual partners | March, 1, 2010 to December, 31,2010
The proportion of people who have intention to be circumcised | March, 1, 2010 to December, 31,2010
The proportion of people who have been circumcised | March, 1, 2010 to December, 31, 2010

CONTACTS AND LOCATIONS:
Overall Officials: Zunyou Wu, MD, PHD, Principal Investigator — National Center for AIDS/STD Control and Prevention, China CDC; Jie Xu, MD, MS, MPH, Principal Investigator — National Center for AIDS/STD Control and Prevention, China CDC
Locations (8):
- China (8):
  - National Center for AIDS/STD Control and Provention, Beijing, Beijing Municipality
  - Center for Disease Control and Prevention, Chongqing City, Chongqing, Chongqing Municipality
  - Center for Disease Control and Prevention,Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - Center for Disease Control and Prevention, Guizhou Province, Guiyang, Guizhou
  - Center for Disease Control and Prevention, Shanghai City, Shanghai, Shanghai Municipality
  - Center for Disease Control and Prevention, Sichuan Province, Chengdu, Sichuan
  - Center for Disease Control and Prevention, Xingjiang Uyghur Autonomous Region, Ürümqi, Xingjiang Uyghur Autonomous Region
  - Center for Disease Control and Prevention, Yunnan Province, Kunming, Yunnan

REFERENCES:
- [Background] Anderson J, Wilson D, Templeton DJ, Grulich A, Carter R, Kaldor J. Cost-effectiveness of adult circumcision in a resource-rich setting for HIV prevention among men who have sex with men. J Infect Dis. 2009 Dec 15;200(12):1803-12. doi: 10.1086/648472. PMID 19909084
- [Background] NIMH Collaborative HIV/STD Prevention Trial Group. The community popular opinion leader HIV prevention programme: conceptual basis and intervention procedures. AIDS. 2007 Apr;21 Suppl 2:S59-68. doi: 10.1097/01.aids.0000266458.49138.fa. PMID 17413265
- [Background] NIMH Collaborative HIV/STD Prevention Trial Group. Formative study conducted in five countries to adapt the community popular opinion leader intervention. AIDS. 2007 Apr;21 Suppl 2:S91-8. doi: 10.1097/01.aids.0000266461.33891.d0. PMID 17413268
- [Background] Feng L, Ding X, Lu R, Liu J, Sy A, Ouyang L, Pan C, Yi H, Liu H, Xu J, Zhao J. High HIV prevalence detected in 2006 and 2007 among men who have sex with men in China's largest municipality: an alarming epidemic in Chongqing, China. J Acquir Immune Defic Syndr. 2009 Sep 1;52(1):79-85. doi: 10.1097/QAI.0b013e3181a4f53e. PMID 19448559
- [Background] Feng LG, Ding XB, Lu RR, Pan CB, Yi HR, Liu HH, Ou YL, Xu J. [HIV prevalence and its associated factors among men who have sex with men in Chongqing]. Zhonghua Yu Fang Yi Xue Za Zhi. 2008 Dec;42(12):870-4. Chinese. PMID 19141218
- [Background] Gao L, Zhang L, Jin Q. Meta-analysis: prevalence of HIV infection and syphilis among MSM in China. Sex Transm Infect. 2009 Sep;85(5):354-8. doi: 10.1136/sti.2008.034702. Epub 2009 Apr 6. PMID 19351623
- [Background] Guo H, Wei JF, Yang H, Huan X, Tsui SK, Zhang C. Rapidly increasing prevalence of HIV and syphilis and HIV-1 subtype characterization among men who have sex with men in Jiangsu, China. Sex Transm Dis. 2009 Feb;36(2):120-5. doi: 10.1097/OLQ.0b013e31818d3fa0. PMID 19125142
- [Background] He Q, Wang Y, Lin P, Raymond HF, Li Y, Yang F, Zhao J, Li J, Ling L, McFarland W. High prevalence of risk behaviour concurrent with links to other high-risk populations: a potentially explosive HIV epidemic among men who have sex with men in Guangzhou, China. Sex Transm Infect. 2009 Sep;85(5):383-90. doi: 10.1136/sti.2009.035808. Epub 2009 Apr 8. PMID 19357129
- [Background] Hong FC, Zhou H, Cai YM, Pan P, Feng TJ, Liu XL, Chen XS. Prevalence of syphilis and HIV infections among men who have sex with men from different settings in Shenzhen, China: implications for HIV/STD surveillance. Sex Transm Infect. 2009 Feb;85(1):42-4. doi: 10.1136/sti.2008.031682. Epub 2008 Jul 24. PMID 18653567
- [Background] Lau JT, Wang M, Tse YK, Gu J, Tsui HY, Zhang Y, Wang N, Cheng F. HIV-related behaviors among men who have sex with men in China: 2005-2006. AIDS Educ Prev. 2009 Aug;21(4):325-39. doi: 10.1521/aeap.2009.21.4.325. PMID 19670968
- [Background] Li L, Cao H, Wu Z, Wu S, Xiao L. Diffusion of positive AIDS care messages among service providers in China. AIDS Educ Prev. 2007 Dec;19(6):511-8. doi: 10.1521/aeap.2007.19.6.511. PMID 18190275
- [Background] Li SW, Zhang XY, Li XX, Wang MJ, Li DL, Ruan YH, Zhang XX, Shao YM. Detection of recent HIV-1 infections among men who have sex with men in Beijing during 2005 - 2006. Chin Med J (Engl). 2008 Jun 20;121(12):1105-8. PMID 18706227
- [Background] Millett GA, Flores SA, Marks G, Reed JB, Herbst JH. Circumcision status and risk of HIV and sexually transmitted infections among men who have sex with men: a meta-analysis. JAMA. 2008 Oct 8;300(14):1674-84. doi: 10.1001/jama.300.14.1674. PMID 18840841
- [Background] Reisen CA, Zea MC, Poppen PJ, Bianchi FT. Male circumcision and HIV status among Latino immigrant MSM in New York City. J LGBT Health Res. 2007;3(4):29-36. doi: 10.1080/15574090802263421. PMID 19002268
- [Background] Ruan S, Yang H, Zhu Y, Ma Y, Li J, Zhao J, McFarland W, Raymond HF. HIV prevalence and correlates of unprotected anal intercourse among men who have sex with men, Jinan, China. AIDS Behav. 2008 May;12(3):469-75. doi: 10.1007/s10461-008-9361-9. Epub 2008 Feb 8. PMID 18259850
- [Background] Ruan Y, Jia Y, Zhang X, Liang H, Li Q, Yang Y, Li D, Zhou Z, Luo F, Shi W, Shao Y. Incidence of HIV-1, syphilis, hepatitis B, and hepatitis C virus infections and predictors associated with retention in a 12-month follow-up study among men who have sex with men in Beijing, China. J Acquir Immune Defic Syndr. 2009 Dec;52(5):604-10. doi: 10.1097/QAI.0b013e3181b31f5c. PMID 19710617
- [Background] Ruan Y, Luo F, Jia Y, Li X, Li Q, Liang H, Zhang X, Li D, Shi W, Freeman JM, Vermund SH, Shao Y. Risk factors for syphilis and prevalence of HIV, hepatitis B and C among men who have sex with men in Beijing, China: implications for HIV prevention. AIDS Behav. 2009 Aug;13(4):663-70. doi: 10.1007/s10461-008-9503-0. Epub 2008 Dec 12. PMID 19082879
- [Background] Ruan Y, Qian HZ, Li D, Shi W, Li Q, Liang H, Yang Y, Luo F, Vermund SH, Shao Y. Willingness to be circumcised for preventing HIV among Chinese men who have sex with men. AIDS Patient Care STDS. 2009 May;23(5):315-21. doi: 10.1089/apc.2008.0199. PMID 19335172
- [Background] Templeton DJ, Millett GA, Grulich AE. Male circumcision to reduce the risk of HIV and sexually transmitted infections among men who have sex with men. Curr Opin Infect Dis. 2010 Feb;23(1):45-52. doi: 10.1097/QCO.0b013e328334e54d. PMID 19935420
- [Background] Xiao Y, Ding X, Li C, Liu J, Sun J, Jia Y. Prevalence and correlates of HIV and syphilis infections among men who have sex with men in Chongqing Municipality, China. Sex Transm Dis. 2009 Oct;36(10):647-56. doi: 10.1097/OLQ.0b013e3181aac23d. PMID 19955876
- [Background] Zhong F, Lin P, Xu H, Wang Y, Wang M, He Q, Fan L, Li Y, Wen F, Liang Y, Raymond HF, Zhao J. Possible increase in HIV and syphilis prevalence among men who have sex with men in Guangzhou, China: results from a respondent-driven sampling survey. AIDS Behav. 2011 Jul;15(5):1058-66. doi: 10.1007/s10461-009-9619-x. PMID 19826942